CLINICAL TRIAL: NCT03373526
Title: Effects of Aerobic Training and Inspiratory Muscle Training in Patients During Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daniel Godoy Martinez (Other)
Responsible Party: Sponsor-Investigator, Daniel Godoy Martinez, PhD, Federal University of Juiz de Fora
Organization: Federal University of Juiz de Fora (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 78682617.9.0000.5133
Record Dates: First submitted 2017-12-05; First posted 2017-12-14 (Actual); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Lymphoma; Myeloma; Leukemia; Aplastic Anemia
Keywords: Hematopoietic Stem Cell Transplantation; Aerobic Exercise; Breathing Exercises; Inspiratory Capacity; Muscle Strength; Exercise Tolerance; Autonomic Nervous System
MeSH Terms: conditions — Lymphoma; Neoplasms, Plasma Cell; Leukemia; Anemia, Aplastic

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, with only statistical analysis blinded
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Physical Training (Active Comparator): Aerobic Training
  Interventions: Other: Aerobic Training
- Combined Physical Training (Experimental): Inspiratory Muscle Training Aerobic Training
  Interventions: Other: Inspiratory Muscle Training; Other: Aerobic Training

INTERVENTIONS:
Other: Inspiratory Muscle Training — The Inspiratory Muscle Training will be perform using using the Power Breathe® device, during 20 minutes daily, five times a week. The protocol will be performed in the sitting position with an established load of 40% of maximal inspiratory pressure.
  Arms: Combined Physical Training
Other: Aerobic Training — The aerobic physical training will be perform using a cycle ergometer, during 20 minutes daily, five times a week, with moderate intensity (50-70% of reserve heart rate).

SUMMARY:
The hospitalization for hematopoietic stem cell transplantation (HSCT) impairs the physical functioning and functional capacity, but aerobic physical training and, more recently, inspiratory muscle training, have shown benefits to patients' health submitted to this intervention. However, is not known the effect of aerobic physical training combined with inspiratory muscle training in hospitalized patients for HSCT. The purpose of the study will be verify the safety, feasibility and effects of the training association.

DETAILED DESCRIPTION:
Sample Patients consecutively admitted to Bone Marrow Transplantation Unit - University Hospital of Juiz de Fora - EBSERH will be included. Patients will be monitored from admission to hospital discharge and randomized by drawing on opaque paper for the Combined Physical Training Group (aerobic physical training + inspiratory muscle training) or the Aerobic Physical Training Group.

Interview Volunteers will go through an interview and directed physical examination. All volunteers will respond to Baecke's questionnaire to investigate habitual physical activity levels.

Feasibility and safety assessment of the study The viability of the study will be verified by: 1) recruitment (recruitment of at least 60% of eligible patients); 2) adherence (achievement of at least 70% of the total number of minutes of the scheduled interventions); 3) friction (percentage of patients who started but did not complete the intervention).

Safety will be verified by the number of spontaneous or unexpected reactions and adverse events resulting from the proposed interventions.

Quality of life and fatigue questionnaire To evaluate the quality of life, the European Organization for Research and Treatment of Cancer (EORTC-Quality of Life Questionnaire-C30) will be used.

The fatigue will be evaluated by the Functional Assessment of Cancer Therapy - Fatigue (FACT-F) questionnaire, validated for the Portuguese language in Brazilian cancer patients.

Anthropometric evaluation Height and body weight will be measured and the BMI calculated.

Evaluation of hematological variables, clinical symptoms, duration of neutropenia and duration of hospital stay Data on hematological variables, the presence of clinical symptoms (diarrhea, constipation, nausea, vomiting, pain and fatigue), duration of neutropenia, need for infusion of red blood cells and platelets, and length of hospital stay in patients' files will be collected and collected.

Evaluation of peripheral muscle strength In order to estimate the muscular strength of lower limbs (LIIII), the sit and stand test will be used for one minute. For the assessment of upper limb muscle strength, the mean value of three maximal hand grip exercises with the dominant limb will be calculated by means of the Jamar® upper limb dynamometer.

Assessment of respiratory muscle strength The maximal inspiratory and expiratory pressures will be measured by digital manovacuometry (MVD300®).

Evaluation of functional capacity The six-minute step test is a simplified functional capacity assessment procedure, often used in the clinical setting because of its ease of execution in the hospital setting. Also, to evaluate the functionality will be applied the Time Up and Go Test.

Assessment of blood pressure and heart rate The oscillometric method will be applied, using the DIXTAL2023® device, which automatically assessing blood pressure. The heart rate will be evaluated continuously by standard derivation of the electrocardiogram cable of the DIXTAL 2023® multiparameter monitor and by the Polar® cardiac frequency meter (model RS800cx).

Evaluation of cardiac autonomic control Cardiac autonomic control will be evaluated by heart rate variability (HRV) analysis.

Evaluation of the cardiac autonomic control profile during hospitalization for HSCT It will be assessed after recording the heart rate for 10 minutes on days of hospital: admission, end of chemotherapy, onset and end of neutropenia and on hospital discharge.

Aerobic physical training protocol All patients admitted to the Bone Marrow Transplantation Unit will participate in the aerobic physical training protocol, as indicated by the Standard Operating Procedure of the Physiotherapy Sector of the Rehabilitation Unit, University Hospital of Juiz de Fora - EBSERH. The aerobic physical training protocol will be performed five times a week, once a day and planned as follows: 1) heating (5-10 minutes), consisting of coordination training and resistance exercises; 2) moderate intensity aerobic physical training (10-20 minutes) performed on a lower limb cycle ergometer; 3) Cooling (5-10 minutes), consisting of muscle stretching and breathing exercises. During the aerobic training, heart rate and peripheral oxygen saturation will be recorded every 2 minutes, as well as blood pressure and subjective effort scale (BORG modified) every 5 minutes. The training target zone will be calculated from 50% to 70% of the reserve heart rate.

Inspiratory Muscle Training Protocol Patients will be familiar with the correct technique for inspiratory muscle training, using the Power Breathe® device, breathing through mouthpiece and nasal clip. Individuals will be instructed to maintain diaphragmatic breathing, respiratory rate between 15 and 20 irpm, during 20 minutes daily, five times a week. The protocol will be performed in the sitting position with an established load of 40% of maximal inspiratory pressure for the combined physical training group.

Clinical safety criteria for contraindication or discontinuation of training protocol The criteria will be to increase the heart rate above 20% of the training target zone, initial systolic blood pressure less than 90 or greater than 160mmHg, blood pressure greater than 170/100 mmHg during exercise, initial oxygen saturation less than 90% or desaturation (greater than 4% during exercise), body temperature greater than 38 °C, severe musculoskeletal pain, chest tightness, major dyspnea or tiredness (greater than 6 on the Borg Scale), dizziness, nausea, vomiting, epistaxis, or any active bleeding, loss or obstruction of the central or peripheral access catheter, loss or obstruction of the bladder catheter / nasogastric/enteral catheter and/or at the patient's request. Moreover, the hemoglobin (less than 7 mg/dl), hematocrit (less than 20%) and platelets (less than 10000 m3) will be absolute contraindications to perform protocols.

Statistical treatment All volunteers included in the study will be evaluated statistically by intention-to-treat analysis. The data collected will first be submitted to exploratory analysis through boxplots, to verify measures of central tendency and dispersion, and to test data normality. From this preliminary investigation will be defined the statistical tests to be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients consecutively admitted to Bone Marrow Transplantation-HU-UFJF-EBSERH for allogeneic or autologous HSCT
* Non-smokers
* Non-alcoholics
* Sedentary for at least three months prior to hospitalization
* Absence of orthopedic limitations and / or cognitive alterations that impede the physical training and the understanding of the evaluation instruments

Exclusion Criteria:

* Patients hospitalized for post-HSCT complications or for other reasons that do not involve HSCT
* Patients who develop metastases and graft-versus-host disease during hospitalization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-11-11 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Inspiratory Pressure Test | On the admission and hospital discharge, an average of 20 to 30 days
  The maximal inspiratory pressure will be measured by digital manovacuometry (cmH20)

SECONDARY OUTCOMES:
Feasibility of Aerobic and Inspiratory Muscle Training | During the entire hospitalization, daily, during an average of 20 to 30 days
  The feasibility of the study will be verified by recruitment (%), adherence (%) and friction (%).
Incidence of Aerobic and Inspiratory Muscle Training - Adverse Events (Safety) | During the entire hospitalization, daily, during an average of 20 to 30 days
  Safety will be verified by the number of spontaneous or unexpected reactions and adverse events resulting from the proposed interventions.
Quality of Life | On the admission and hospital discharge, an average of 20 to 30 days
  To evaluate the quality of life, the European Organization for Research and Treatment of Cancer (EORTC-QLQ-C30) will be used. It will be considered the score of the global health, functional health and symptoms domains.
Fatigue | On the admission and hospital discharge, an average of 20 to 30 days
  The fatigue will be evaluated by the total score of Functional Assessment of Cancer Therapy - Fatigue (FACT-F) questionnaire.
Hematological Variables | During the entire hospitalization, daily, during an average of 20 to 30 days
  Patient records will be consulted and collected daily in order to verify the white cells, red cells and platelets counts.
Clinical Symptoms | During the entire hospitalization, daily, during an average of 20 to 30 days
  Patient records will be consulted and collected daily in order to verify the presence of diarrhea, pain, nausea, vomiting, fever, hair loss, fatigue, shortness of breath.
Duration of Neutropenia | During the entire hospitalization, daily, during an average of 20 to 30 days
  Patient records will be consulted and collected daily in order to verify the number of the days in which the patient will be in neutropenia.
Duration of Hospitalization | During the entire hospitalization, daily, during an average of 20 to 30 days
  Patient records will be consulted and collected daily in order to verify the number of the days in which the patient will be hospitalized.
Muscle Strength of Lower Limbs | On the admission and hospital discharge, an average of 20 to 30 days
  The muscular strength of lower limbs (LIIII) will be verified by the sit and stand test will be used for one minute (number of repetitions).
Muscle Strength of Upper Limbs | On the admission and hospital discharge, an average of 20 to 30 days
  For the assessment of upper limb muscle strength will be used Jamar® upper limb dynamometer (kgf).
Functional Capacity | On the admission and hospital discharge, an average of 20 to 30 days
  The six-minute step test will be used and the number of up and down steps will be considered.
Functionality | On the admission and hospital discharge, an average of 20 to 30 days
  The Time Up and Go Test will be used and the time to execute the test will be considered in seconds (s).
Blood Pressure | During the entire hospitalization, daily, during an average of 20 to 30 days
  The oscillometric method will be applied, using the DIXTAL2023® device to evaluate the systolic, diastolic and mean blood pressure (mmHg).
Heart Rate | During the entire hospitalization, daily, during an average of 20 to 30 days
  The heart rate (beats per minute) will be evaluated continuously by standard derivation of the electrocardiogram cable of the DIXTAL 2023® multiparameter monitor and by the Polar® cardiac frequency meter (model RS800cx).
Cardiac Autonomic Control | Hospital admission day, the end of chemotherapy day, the beginning and end of neutropenia days and the day of hospital discharge, during an average of 20 to 30 days to study completion.
  The cardiac autonomic control will be assessed by the frequency (ms2 and nu) and time domains (ms) of heart rate variability analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel G Martinez, PhD, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- University Hospital-EBSERH, Juiz de Fora, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brooks D, Solway S, Gibbons WJ. ATS statement on six-minute walk test. Am J Respir Crit Care Med. 2003 May 1;167(9):1287. doi: 10.1164/ajrccm.167.9.950. No abstract available. PMID 12714344
- [Background] Bargi G, Guclu MB, Aribas Z, Aki SZ, Sucak GT. Inspiratory muscle training in allogeneic hematopoietic stem cell transplantation recipients: a randomized controlled trial. Support Care Cancer. 2016 Feb;24(2):647-659. doi: 10.1007/s00520-015-2825-3. Epub 2015 Jul 2. PMID 26135532
- [Background] da Costa CH, da Silva KM, Maiworm A, Raphael Y, Parnayba J, Da Cal M, Figueira B, Condesso D, Rufino R. Can we use the 6-minute step test instead of the 6-minute walking test? An observational study. Physiotherapy. 2017 Mar;103(1):48-52. doi: 10.1016/j.physio.2015.11.003. Epub 2015 Dec 14. PMID 27012823
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210
- [Background] Poreba M, Poreba R, Gac P, Usnarska-Zubkiewicz L, Pilecki W, Piotrowicz E, Piotrowicz R, Rusiecki L, Kuliczkowski K, Mazur G, Sobieszczanska M. Heart rate variability and heart rate turbulence in patients with hematologic malignancies subjected to high-dose chemotherapy in the course of hematopoietic stem cell transplantation. Ann Noninvasive Electrocardiol. 2014 Mar;19(2):157-65. doi: 10.1111/anec.12108. Epub 2013 Nov 8. PMID 24206437
- [Background] Wood WA, Deal AM, Reeve BB, Abernethy AP, Basch E, Mitchell SA, Shatten C, Hie Kim Y, Whitley J, Serody JS, Shea T, Battaglini C. Cardiopulmonary fitness in patients undergoing hematopoietic SCT: a pilot study. Bone Marrow Transplant. 2013 Oct;48(10):1342-9. doi: 10.1038/bmt.2013.58. Epub 2013 Apr 15. PMID 23584437
- [Derived] Almeida LB, Laterza MC, Rondon MUPB, de Matos LDNJ, Granger CL, Denehy L, Oliveira CC, Trevizan PF, Martinez DG. Inspiratory muscle training in addition to conventional physical rehabilitation in hospitalized patients undergoing hematopoietic stem cell transplantation: a randomized controlled trial. Support Care Cancer. 2022 Nov;30(11):9393-9402. doi: 10.1007/s00520-022-07373-z. Epub 2022 Sep 29. PMID 36173561
- [Derived] de Almeida LB, Trevizan PF, Laterza MC, Hallack Neto AE, Perrone ACASJ, Martinez DG. Safety and feasibility of inspiratory muscle training for hospitalized patients undergoing hematopoietic stem cell transplantation: a randomized controlled study. Support Care Cancer. 2020 Aug;28(8):3627-3635. doi: 10.1007/s00520-019-05209-x. Epub 2019 Dec 5. PMID 31807987